CLINICAL TRIAL: NCT04810260
Title: Implementing, Validating, and Disseminating a Patient-facing Mobile Health Application for HIV Infected and Uninfected Women With Co-morbid Conditions in the Outpatient Setting
Brief Title: Implementing, a Mobile Health Application for HIV Infected and Uninfected Women With Co-morbidities in the Outpatient Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Sunit P. Jariwala, Associate Profesor, Montefiore Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-12608
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Mobile Health; Asthma; Diabetes Mellitus
Keywords: mobile health; asthma; diabetes mellitus
MeSH Terms: conditions — Asthma; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV + (Active Comparator): Patients will have the application and use it to increase their awareness about their medical condition.
  Interventions: Behavioral: Use mobile health app (WellXcel) to increase knowledge
- HIV - (Active Comparator): Patients will have the application and use it to increase their awareness about their medical condition.
  Interventions: Behavioral: Use mobile health app (WellXcel) to increase knowledge

INTERVENTIONS:
Behavioral: Use mobile health app (WellXcel) to increase knowledge — Download the app (WellXcel) to the mobile device

SUMMARY:
This is a pilot study conducted at the Bronx MWCCS Clinical Research Site in the Bronx, NY.

We will recruit 60 individuals with coexisting asthma and/or Type 2 DM from this cohort.

During the 3 month study period, these 60 participants will receive a comprehensive mobile health (mHealth) app, WELLXcel which includes: 1) guideline-based asthma and diabetes education delivered through interactive features such as animated videos and tailored push notifications; 2) the collection of PRO measures to enable patients symptom self-tracking.

During this study, we will evaluate the association between baseline digital health literacy and favorable clinical outcomes related to the WELLXcel study intervention.

DETAILED DESCRIPTION:
The study objectives and hypotheses are:

Objective 1. To adapt (including a single platform for multiple chronic conditions) and refine WELLXcel for adult women with and without HIV. Hypothesis 1: WELLXcel will be associated with a high level of adoption and will be successfully refined based on patient feedback. Objective 2. To conduct a pilot study to assess the impact of the adapted and refined WELLXcel program on clinical and process outcomes among women with and without HIV.

Hypothesis 2: WELLXcel will be associated with a high level of patient satisfaction and usage, improved asthma and diabetes knowledge, improvements in health quality of life, and improved self-reported asthma control and diabetes related quality of life compared to usual care. Primary outcomes: Asthma control measured by the Asthma Control Test (ACT) and diabetes quality of life measured by the Diabetes Quality of Life (DQOL) instrument.

Secondary outcomes: Process outcomes - patient satisfaction regarding the WELLXcel intervention measured by the validated Questionnaire for User Interface Satisfaction (QUIS) and the Unified Theory of Acceptance and Use of Technology (UTAUT) questionnaire; patient usage of WELLXcel as determined by Google Analytics (integrated within the WELLXcel app) and the WELLXcel backend administrative panel; asthma knowledge (measured by the Asthma Illness Representation Scale and diabetes knowledge (measured by the Diabetes Knowledge Questionnaire-24)[24] ; diabetes self-management and self-efficacy as measured by the Diabetes Self-Management Questionnaire (DSMQ) and Diabetes Empowerment Scale-Short Form (DES-SF), respectively. Clinical outcomes - Asthma quality of life measured by the Mini-Asthma Quality of Life Questionnaire (mini- AQLQ); asthma and/or diabetes related emergency department visits and hospitalizations; and the Patient Health Questionnaire-9 (PHQ-9) for depression.

Subjects:

Inclusion Criteria: English-speaking women >18 years with: (a) persistent asthma (diagnosis via self-report) on a daily controller medication and/or Type 2 diabetes mellitus (diagnosis via self-report) on at least one oral hypoglycemic medication and/or Insulin; (b) able to give informed consent; and (c) Smartphone (iOS or Android) access. Exclusion Criteria: (a) use of oral corticosteroids in the 2 weeks prior to the baseline visit; (b) pregnancy; (c) chronic illness with organ failure (heart failure, severe liver disease, chronic kidney disease stage 3-4 or dialysis) or requiring chemotherapy or steroid use; (d) severe psychiatric or cognitive problems that would prohibit an individual from understanding and completing the protocol; and (e) patients that previously received the ASTHMAXcel application.

Investigators will recruit 30 HIV infected and 30 HIV uninfected adult women with persistent asthma and/or Type 2 DM and fulfilling the study's inclusion criteria from the MWCCS cohort. At each study site, patients will be prescreened for eligibility using data from WIHS (Women's Interagency HIV Study) to identify those who meet the inclusion criteria. In adapting with the ongoing COVID-19 pandemic and our existing AHRQ study protocols, patient recruitment and study sessions will be conducted virtually to support physical distancing and reduce the risk of contracting and transmitting COVID- 19 infection. The study coordinators will call potential participants to describe the study and obtain voluntary informed consent from interested patients.

Regarding the consent process, the study participant may choose to complete the e-consent (as a form administered through our project's REDCap database via an e-mail link sent to the patients who will read and electronically sign the consent) or verbal consent (the consent will be read out to the patients who will subsequently provide verbal confirmation of having understood the consent text and affirm consenting to the study).

Voluntary informed consent will include a discussion of the study purpose, study procedures, research virtual visit schedule, reimbursement, confidentiality of research records, and risks, benefits, and alternatives to study participation. Investigators will discuss that research participation is voluntary, and participants will be notified that they can discontinue participation at any time.

The study coordinator will document that the purpose, risks, benefits, and alternative treatments were explained to the participant, that the participant agreed to participate in this protocol, and the date and time consent was obtained. A copy of the HIPAA form and a copy of the informed consent document will be given to the participant. In either case, whether the e-consent or the verbal consent form is obtained, the participant will receive the consent document, which will be printed and mailed out to them. All informed consent and HIPAA documents will be submitted to, and approved by, the Albert Einstein College of Medicine IRB. E-consent forms will be stored within our project's secure REDCap database.

Sixty patients who provide voluntary informed consent will be invited to the remotely conducted (via Zoom) baseline visit, which consists of downloading the app to the patient's smartphone, explaining the app's functionality, having the patients complete the WELLXcel animated educational videos and baseline questionnaires administered by REDCap. Assessments will be conducted at baseline followed by 1, 2, and 3 months after baseline. The baseline survey and the subsequent assessments will include process outcomes (patient usage, acceptance and satisfaction with the app) as well as measures of disease morbidity (asthma and diabetes control, utilization measures in terms of asthma and/or diabetes-related ED visits and hospitalizations) and quality of life questionnaires. Based on our preliminary studies, patients with 1 condition will take approximately 20 minutes to complete the surveys during a given study visit. Patients with 2 conditions will take approximately 45 minutes to complete the surveys. Each study visit will also include brief semi-structured interviews to gather patient feedback (e.g. problems with using the app). Investigators will also use the Google Analytics and WELLXcel admin panel to evaluate app usage patterns and click-through data to better understand how the app is used, which may lead to the identification of additional usability pitfalls. Investigators will use our existing REDCap project database to store app-collected data and responses to REDCap-administered questionnaires. At the 2 month visit, we will conduct exit interviews with each study participant to enable us to refine the app for our upcoming studies.

To assess digital health literacy and concurrently validate our digital health literacy tool, the study baseline session will also include NVS, eHEALS, and our digital health literacy tool. At the subsequent 1-month assessment, digital health literacy tool will be re-administered to evaluate test-retest reliability. There is no previously defined cut-off score on the eHEALS questionnaire which simply defines a patient as eHealth literate' or 'not eHealth literate'. For this study, investigators will define literacy as follows: a score of 32 or higher (out of a 40 point maximum score) will indicate 'good EHL', a score of 24-31 will indicate 'moderate EHL', and a score below 24 will indicate 'low EHL'. On the objective digital health literacy tool, 'good EHL' will be defined as a score from 8-10 (out of a maximum of 10), a score of 5-7 will indicate 'moderate EHL', and a score below 5 will indicate 'low EHL'. Patients will complete all health literacy questionnaires via REDCAP generated e-mail survey links during the study sessions.

ELIGIBILITY:
Inclusion Criteria:

English-speaking women >18 years with:

* persistent asthma (diagnosis via self-report) on a daily controller medication and/or Type 2 diabetes mellitus (diagnosis via self-report) on at least one oral hypoglycemic medication and/or Insulin;
* able to give informed consent;
* Smartphone (iOS or Android) access.

Exclusion Criteria:

* use of oral corticosteroids in the 2 weeks prior to the baseline visit;
* pregnancy
* chronic illness with organ failure (heart failure, severe liver disease, chronic kidney disease stage 3-4 or dialysis) or requiring chemotherapy or steroid use;
* severe psychiatric or cognitive problems that would prohibit an individual from understanding and completing the protocol;
* patients that previously received the ASTHMAXcel application.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological woman
Enrollment: 42 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Asthma control measured by the Asthma Control Test. | 1 month
  Surveys will be applied.
Asthma control measured by the Asthma Control Test. | 2 months
  Surveys will be applied.
Asthma control measured by the Asthma Control Test. | 3 months
  Surveys will be applied.
Diabetes quality of life measured by the Diabetes Quality of Life instrument | 1 month
  Surveys will be applied.
Diabetes quality of life measured by the Diabetes Quality of Life instrument | 2 months
  Surveys will be applied.
Diabetes quality of life measured by the Diabetes Quality of Life instrument | 3 months
  Surveys will be applied.

SECONDARY OUTCOMES:
patient satisfaction regarding the WELLXcel intervention measured by the validated Questionnaire for User Interface Satisfaction (QUIS) | 1 month
  Surveys will be applied
patient satisfaction regarding the WELLXcel intervention measured by the validated Questionnaire for User Interface Satisfaction (QUIS) | 2 months
  Surveys will be applied
patient satisfaction regarding the WELLXcel intervention measured by the validated Questionnaire for User Interface Satisfaction (QUIS) | 3 months
  Surveys will be applied
Unified Theory of Acceptance and Use of Technology questionnaire | 1 months
  Surveys will be applied
Unified Theory of Acceptance and Use of Technology questionnaire | 2 months
  Surveys will be applied
Unified Theory of Acceptance and Use of Technology questionnaire | 3 months
  Surveys will be applied
Patient usage of WELLXcel from the backend administrative panel. | 1 month
  Analyse the administrative panel.
Patient usage of WELLXcel from the backend administrative panel. | 2 months
  Analyse the administrative panel.
Patient usage of WELLXcel from the backend administrative panel. | 3 months
  Analyse the administrative panel.
Diabetes self-management and self-efficacy as measured by the Diabetes Self-Management Questionnaire | 1 months
  Surveys will be applied
Diabetes self-management and self-efficacy as measured by the Diabetes Self-Management Questionnaire | 2 months
  Surveys will be applied
Diabetes self-management and self-efficacy as measured by the Diabetes Self-Management Questionnaire | 3 months
  Surveys will be applied
Diabetes Empowerment Scale-Short Form | 1 months
  Surveys will be applied
Diabetes Empowerment Scale-Short Form | 2 months
  Surveys will be applied
Diabetes Empowerment Scale-Short Form | 3 months
  Surveys will be applied
Asthma quality of life measured by the Mini-Asthma Quality of Life Questionnaire. | 1 months
  Surveys will be applied
Asthma quality of life measured by the Mini-Asthma Quality of Life Questionnaire. | 2 months
  Surveys will be applied
Asthma quality of life measured by the Mini-Asthma Quality of Life Questionnaire. | 3 months
  Surveys will be applied
Asthma and/or diabetes related emergency department visits and hospitalizations | 1 month
  Patient reports will be used.
Asthma and/or diabetes related emergency department visits and hospitalizations | 2 months
  Patient reports will be used.
Asthma and/or diabetes related emergency department visits and hospitalizations | 3 months
  Patient reports will be used.
Patient Health Questionnaire-9 for depression | 1 month
  Surveys will be applied
Patient Health Questionnaire-9 for depression | 2 months
  Surveys will be applied
Patient Health Questionnaire-9 for depression | 3 months
  Surveys will be applied

CONTACTS AND LOCATIONS:
Overall Officials: Sunit Jariwala, MD, Principal Investigator — Albert Einstein College of Medicine/Montefiore MC
Locations (1):
- Albert Einstein College Of Medicine/Montefiore MC, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
Only study coordinators and research assistants will have the data.

REFERENCES:
- [Background] Gingo MR, Wenzel SE, Steele C, Kessinger CJ, Lucht L, Lawther T, Busch M, Hillenbrand ME, Weinman R, Slivka WA, McMahon DK, Zhang Y, Sciurba FC, Morris A. Asthma diagnosis and airway bronchodilator response in HIV-infected patients. J Allergy Clin Immunol. 2012 Mar;129(3):708-714.e8. doi: 10.1016/j.jaci.2011.11.015. Epub 2011 Dec 15. PMID 22177327
- [Background] Kendall CE, Wong J, Taljaard M, Glazier RH, Hogg W, Younger J, Manuel DG. A cross-sectional, population-based study measuring comorbidity among people living with HIV in Ontario. BMC Public Health. 2014 Feb 13;14:161. doi: 10.1186/1471-2458-14-161. PMID 24524286
- [Background] Petoumenos K, Huang R, Hoy J, Bloch M, Templeton DJ, Baker D, Giles M, Law MG, Cooper DA. Prevalence of self-reported comorbidities in HIV positive and HIV negative men who have sex with men over 55 years-The Australian Positive & Peers Longevity Evaluation Study (APPLES). PLoS One. 2017 Sep 8;12(9):e0184583. doi: 10.1371/journal.pone.0184583. eCollection 2017. PMID 28886173
- [Background] Richtering SS, Morris R, Soh SE, Barker A, Bampi F, Neubeck L, Coorey G, Mulley J, Chalmers J, Usherwood T, Peiris D, Chow CK, Redfern J. Examination of an eHealth literacy scale and a health literacy scale in a population with moderate to high cardiovascular risk: Rasch analyses. PLoS One. 2017 Apr 27;12(4):e0175372. doi: 10.1371/journal.pone.0175372. eCollection 2017. PMID 28448497
- [Background] Nguyen J, Moorhouse M, Curbow B, Christie J, Walsh-Childers K, Islam S. Construct Validity of the eHealth Literacy Scale (eHEALS) Among Two Adult Populations: A Rasch Analysis. JMIR Public Health Surveill. 2016 May 20;2(1):e24. doi: 10.2196/publichealth.4967. PMID 27244771

DOCUMENTS (1):
  • Informed Consent Form (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT04810260/ICF_000.pdf